CLINICAL TRIAL: NCT06698458
Title: A Study to Assess the Safety of Intratumoral Diffusing Alpha Radiation Emitters With Chemotherapy for the Treatment of Locally Advanced and Metastatic Pancreatic Cancer
Brief Title: Alpha Radiation Emitters Device for the Treatment of Pancreatic Cancer With Chemotherapy for the Treatment of Locally Advanced and Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-PANC-09
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma; Metastatic Pancreatic Cancer
Keywords: Alpha radiation; pancreatic cancer; Pancreatic Adenocarcinoma; Unresectable Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 15 patients in each cohort for a total of 30 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Patients with locally advanced pancreatic adenocarcinoma (Experimental): Patients will begin mFOLFIRINOX treatment and will undergo DaRT placement during the first 4 cycles. Follow-up will continue up to 6 months after enrollment.
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)
- Patients with metastatic pancreatic adenocarcinoma (Experimental): Patients will begin mFOLFIRINOX treatment and will undergo DaRT placement during the first 4 cycles. Follow-up will continue up to 6 months after enrollment.
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — DaRT source will be inserted using endoscopy into the tumor. The sources release by recoil into the tumor short-lived alpha-emitting atoms
  Other Names: DaRT

SUMMARY:
This is a multi-center clinical study enrolling up to 30 participants (15 patients in each cohort). The primary objective of the study is to evaluate the safety of Alpha DaRT in combination with chemotherapy, based on the cumulative incidence rate, severity and outcome of device related AEs. Classification of AEs will be done according to CTCAE V5. The secondary objectives of the study are to:

* Assess efficacy of the Alpha DaRT sources in combination with chemotherapy, determined by overall and progression-free survival.
* Assess pain control
* Assess rate of surgical resection in Cohort 1.

DETAILED DESCRIPTION:
This study will be a prospective, interventional, open label, two cohort, multiple center study to assess the efficacy of Alpha DaRT in combination with chemotherapy. Eligible patients with newly diagnosed pancreatic cancer will be categorized into one of the following two cohorts according to their disease state at baseline:

1. Locally advanced
2. Metastatic. Patients will begin mFOLFIRINOX treatment and will undergo DaRT placement during the first 4 cycles. Follow-up will continue up to 6 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically proven newly diagnosed locally advanced inoperable pancreatic adenocarcinoma (Cohort 1) OR histologically and/or cytologically proven newly diagnosed metastatic pancreatic adenocarcinoma (Cohort 2).
* Patients will start treatment with mFOLFIRINOX (up to 4 cycles) before DaRT insertion
* Target lesion is technically amenable for Alpha DaRT sources implantation.
* Measurable lesion per RECIST (version 1.1) criteria
* Lesion size ≤ 5 cm in the longest diameter
* Interstitial radiation indication validated by a multidisciplinary team.
* ECOG Performance Status Scale 0 -2
* Life expectancy is more than 6 months
* WBC ≥ 3500/μl, granulocyte ≥ 1500/μl
* Platelet count ≥60,000/μl
* Creatinine ≤1.9 mg/dL
* AST and ALT ≤ 2.5 X upper limit of normal (ULN)
* INR < 1.4 for patients not on Warfarin
* Age ≥18 years old
* Subjects are willing and able to sign an informed consent form
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test before the Ra-224 implantation and are required to use an acceptable contraceptive method to prevent pregnancy for 3 months after initiation of Alpha DaRT therapy.
* Patients must agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after DaRT insertion.

Exclusion Criteria:

* For Cohort 1 only: Borderline unresectable pancreatic cancer, and/or fit for surgical exploration unless patient refuses surgery.
* For Cohort 1 and Cohort 2: Prior treatment for pancreatic cancer, including chemotherapy except for 1 - 4 cycles of mFOLFIRINOX, radiation therapy, immunotherapy, etc.
* Known hypersensitivity to any of the components of the treatment.
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids.
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial or interfere with the study endpoints.
* Has a known additional malignancy that is progressing or requires active treatment.

Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, low risk prostate cancer, or in situ cervical cancer.

* Patient requires treatment not specified in this protocol which may conflict with the endpoints of this study including evaluation of response or toxicity of DaRT.
* Patients do not agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after DaRT insertion.
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator).
* Breastfeeding women or women of childbearing potential unwilling or unable to use an acceptable contraceptive method to prevent pregnancy for 3 months after DaRT insertion
* Patients who are at high risk of complications from radiation due to genetic conditions/mutations, inflammatory bowel disease, or connective tissue disease.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety -Serious adverse events | From Day 0 ,up to 24 months.
  The primary endpoint is the incidence of treatment-related Serious Adverse Events (SAEs) graded according to CTCAE v5.0

SECONDARY OUTCOMES:
Complete or pain response | 30 days and 2 months post-procedure
  Complete or partial pain response at 30 days and 2 months postprocedure as compared to baseline based on average pain scale using BPI-SF (Brief Pain Inventory - Short Form) used to evaluate the severity of a patient's pain, 0-no pain, 1 to 3- mild pain, 4 to 7- moderate pain, 8 to 10- severe pain .
Percentage of locally advanced that became surgically resectable | 6 and 24 months
  For cohort 1 only: Percentage of locally advanced patients with tumors that became surgically resectable after DaRT treatment

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Goodyear, Arizona
  - Honor Health, Scottsdale, Arizona
  - Cedars-Sinai, Los Angeles, California
  - Advent Health Cancer Institute, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Bassett Healthcare Network, Cooperstown, New York
  - NYU Langone Health, New York, New York
  - Lenox hill Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Texas Oncology, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University Cancer and Diagnostic, Houston, Texas
- Jewish General Hospital, Montreal, Quebec, Canada
- Hadassah Ein Kerem, Jerusalem, Israel